CLINICAL TRIAL: NCT00524602
Title: A Nonrandomized Observertionel Study That Will Show the Utility and the Safety by Using the Remote Magnetic Navigation of Ablationcatheters and the Stereotaxis Equipment
Brief Title: The Use of Remote Magnetic Navigation in Catheter Ablation of Heart Arrythmia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Jesper Hastrup Svendsen, Rigshospitalet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STEREOTAXIS study; No funding
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2007-08

CONDITIONS: Arrythmia
Keywords: Stereotaxis; Arrythmia; Catheter ablation; Heart
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Catheter ablation using the Stereotaxis equipment — Energy delivery through ablation catheter during an interventional catheterisation of the heart.
  Other Names: Radiofrequency ablation

SUMMARY:
Patients with several heart arrythmia can potentially be cured by catheterablation. For some arrythmias 95% of the patients are cured. Also patients with atrial fibrillation are cured by catherablation even though the effect is not as impressive as for other cardiac arrythmias. About 70% of patients with paroxystic and persistant atrial fibrillation are cured. Most of the remaining obtain a reduction of their symptoms.

At conventional ablation of atrial fibrillation the catheters are manually navigated to the ideal anatomic position where to isolate the pulmonary veins from the left atrium.

Lately it has been possible to navigate the ablationcatheters using 'remote magnetic navigation' using a magnetic based navigation equipment, Stereotaxis.

The Heartcentre of Rigshospitalet had this Stereotaxis equipment installed in the autumn of 2006.

We will investigate the utility and safety of using this remote magnetic navigation/Stereotaxis.

DETAILED DESCRIPTION:
The purpose on this study is to show the utility and the safety by using the remote magnetic navigation of ablation catheters with the Stereotaxis equipment at ablations of

* atrial fibrillation, atrial flutter and other arrythmias
* childrens arrythmias
* arrythmias of patients with pacemaker or ICD (Implantable Cardiac Defibrillator)

ELIGIBILITY:
Inclusion Criteria:following patients that need catheter ablation:

* Patients with atrial fibrillation
* Patients with artial flutter
* Patients with other tachy arrythmia
* Patients with paceaker/ICD

Exclusion Criteria:

* Patients with anamnestic psycosis or other conditions where information is impossible or insure to give
* Contraindication to magnetic ablation therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2007-06; Primary Completion 2012-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Clinical effect and safety of ablation | 3 month after procedure
  Stroke and death

SECONDARY OUTCOMES:
Feasibility of remote navigation | within 3 months
  Succesrate

CONTACTS AND LOCATIONS:
Overall Officials: Xu Chen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark